CLINICAL TRIAL: NCT02955914
Title: The Effect of Patient Optimism & Pessimism on Recovery From Elective Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr Vikki Hughes (Other Government)
Responsible Party: Sponsor-Investigator, Dr Vikki Hughes, Senior R&D Manager, Papworth Hospital NHS Foundation Trust
Organization: Papworth Hospital NHS Foundation Trust (Other Government)
Other Study IDs: P02022
Record Dates: First submitted 2016-09-15; First posted 2016-11-04 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Mental Stress
Keywords: Optimism; Pessimism; Recovery; Elective Cardiac surgery
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Optimism: Based on quality of life assessment
- Pessimism: Based on quality of life assessment

SUMMARY:
Before a heart operation, patient outlook may be either pessimistic or optimistic. Previous research on this topic has focused on patient reported quality of life but has never examined measurable clinical outcomes such as length of hospital stay.This pilot study hopes to establish whether patient outlook (optimistic or pessimistic) before a heart operation can influence recovery and length of hospital stay. If there is a difference, then a case can be made for providing psychological support before an operation in the hope of modifying outlook and thus improving patient care and reducing hospital stay and NHS costs. Patients will be recruited over a 12month period. Their outlook (pessimistic or optimistic) will be ascertained using two standardised questionnaires. Their recovery and length of stay will be recorded. The study will answer the research question and determine whether outlook has an impact on recovery. Depending on the results, this study could provide opportunities for additional future research into modifying outlook with a view to improving patient care and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Elective planned cardiac surgery
* Consent to participate

Exclusion Criteria:

* Patients diagnosed with clinical depression
* Patients deemed not competent to provide consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be elective cardiac surgical patients undergoing major cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Discharge from hospital (average of 10 days)

SECONDARY OUTCOMES:
Length of ITU stay | 2 days
Risk-adjusted survival | Discharge from hospital (average of 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Mills, Principal Investigator — Papworth Hospital NHS
Locations (1):
- Papworth Hospital NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data will be disseminated among the research team. Patients can see a copy of the final report upon request.